CLINICAL TRIAL: NCT01033097
Title: A Multicenter, Randomized, Double-blinded, Placebo and Positive Controlled Study to Evaluate the Anti-pruritic Effect, Safety and Tolerability, Systemic and Skin Exposure, After 2 Weeks of Treatment With a Microemulsion Formulation of DNK333 in Atopic Dermatitis Patients
Brief Title: Safety and Efficacy of DNK333 in Atopic Dermatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDNK333B2103; EudraCT 2009-012098-36 (Other: EMEA)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Pruritus in Patients With Atopic Dermatitis
Keywords: Dermatitis; inflammatory skin disease; itch; eczema
MeSH Terms: conditions — Dermatitis; Pruritus; Eczema | interventions — DNK 333; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (9):
- DNK333 5 mg (Experimental)
  Interventions: Drug: DNK333 5 mg
- Placebo to DNK333 5mg (Placebo Comparator)
  Interventions: Drug: Placebo to 5 mg
- DNK333 25 mg (Experimental)
  Interventions: Drug: DNK333 25 mg
- Placebo to DNK333 25 mg (Placebo Comparator)
  Interventions: Drug: Placebo to 25 mg
- DNK333 100 mg (Experimental)
  Interventions: Drug: DNK333 100 mg
- Placebo to DNK333 100 mg (Placebo Comparator)
  Interventions: Drug: Placebo to 100 mg
- Betamethasone 4 mg (Active Comparator)
  Interventions: Drug: Betamethasone 4 mg
- DNK333 1 mg (Experimental)
  Interventions: Drug: DNK333 1mg
- placebo 1mg (Placebo Comparator)
  Interventions: Drug: Placebo to 1mg

INTERVENTIONS:
Drug: DNK333 5 mg — 5 mg oral
  Arms: DNK333 5 mg
Drug: Placebo to 5 mg — 5 mg placebo oral
  Arms: Placebo to DNK333 5mg
Drug: DNK333 25 mg — 25 mg oral
  Arms: DNK333 25 mg
Drug: Placebo to 25 mg — 25 mg placebo oral
  Arms: Placebo to DNK333 25 mg
Drug: DNK333 100 mg — 100 mg oral
  Arms: DNK333 100 mg
Drug: Placebo to 100 mg — 100 mg placebo oral
  Arms: Placebo to DNK333 100 mg
Drug: Betamethasone 4 mg — 4 mg oral
  Arms: Betamethasone 4 mg
Drug: DNK333 1mg — 1 mg oral
  Arms: DNK333 1 mg
Drug: Placebo to 1mg — 1 mg placebo oral
  Arms: placebo 1mg

SUMMARY:
This study will assess the safety and efficacy of DNK333 in patients with atopic dermatitis suffering from pruritus, who require systemic treatment of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female atopic dermatitis patients,18 to 60 years of age inclusive, who fulfill the following criteria:
* Requirement of systemic therapy
* Itch VAS score higher than 50 mm
* EASI score higher than 8

Exclusion Criteria:

* Women of child-bearing potential who are not willing to use two highly effective methods of contraception are not allowed in the study. Similarly, men who are not willing to use two acceptable methods of contraception are not allowed in the study.
* Any systemic immunosuppressive treatment and/or phototherapy within 4 weeks prior to the first dosing.
* Use of any systemic antihistamines or topical corticosteroids within one week prior to first dosing and for the duration of the treatment period. Any other topical or oral treatment for atopic dermatitis (except emollients prescribed by the investigator) within 2 weeks prior to the first dosing will also be excluded.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of DNK333 in reduction in pruritus in atopic dermatitis patients, as measured by actigraphy and visual analogue scale (VAS) | 2 weeks

SECONDARY OUTCOMES:
Evaluate the therapeutic benefit from the patient's perspective of DNK333 to reduce pruritus as assessed by the Patient Benefit Index for Pruritus (PBIfP) | 2 weeks
Efficacy of DNK333 to reduce dermatitis as measured by the atopic dermatitis score and the Eczema Severity Index (EASI) | 2 weeks
Safety and tolerability of DNK333 in atopic dermatitis patients | 2 weeks
the plasma pharmacokinetics and skin exposure following treatment of atopic dermatitis patients with DNK333. | 2 weeks
Assess the health-related quality of life by using the Quality of Life for Atopic Dermatitis (QoLIAD) score. | 2 weeks
Compare the pharmacokinetics of DNK333 administered as an oral microemulsion drinking solution to a solid dispersion tablet in steady state. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigator Site, Hanover
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster